CLINICAL TRIAL: NCT05699265
Title: Cardiovasculorenal Phenotyping in Fabry Disease Through Noninvasive Testing
Acronym: VDFP
Status: Terminated | Type: Observational
Why Stopped: The sponsor withdrew funding since there was no progress with this study for a significant amount of time.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-0779 VDFP
Record Dates: First submitted 2023-01-12; First posted 2023-01-26 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — Blood Pressure Monitoring, Ambulatory; Exercise Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Fabry Disease Follow-Up Patients
  Interventions: Diagnostic Test: Measures of arterial stiffness and endothelial function; Diagnostic Test: Ambulatory blood pressure monitoring; Diagnostic Test: Cardiopulmonary exercise testing (CPET); Diagnostic Test: Serum and urine biomarkers

INTERVENTIONS:
Diagnostic Test: Measures of arterial stiffness and endothelial function — baseline cMRI, vascular reactivity studies, and CPET
Diagnostic Test: Ambulatory blood pressure monitoring — A manual blood pressure with a mercury sphygmomanometer will be performed in order to have an accurate baseline measurement. The SphygmoCor SCOR-PVx System (Atcor Medical, Syndey, Australia), previously validated in the young, will be used for the assessment of PWV (pulse wave velocity) and the Heart Rate Variability (HRV).
Diagnostic Test: Cardiopulmonary exercise testing (CPET) — Cardiopulmonary exercise testing will be performed, and the patients will have a baseline oxygen uptake at rest to determine the rates for testing. A 12 lead ECG, heart rate, a 12 lead rhythm strip, and a 6 lead rhythm strip will be recorded. Oxygen consumption and carbon dioxide production will be measured. Blood pressure will be measured. Perceived exertion will be obtained during each workload using the Borg Scale. The results for submaximal effort testing will be derived from completed maximal testing. The outcome measures will be obtained once the subject reaches anaerobic threshold.
Diagnostic Test: Serum and urine biomarkers — Clinical labs drawn will include plasma and urine globotriaosylsphingosine (lyso-Gb3), globotriaosylceramide (GL3), blood urea nitrogen, creatinine, cystatin C, urinalysis, urine protein, urine microalbumin and urine creatinine. Labs specific for this study will include N-acetyl-β-glucosaminidase, urine neutrophil gelatinase-associated lipocalin (NGAL), and kidney injury molecule 1 (KIM-1). All data will be obtained at three different time intervals: enrollment, 1 year and 2 years.

SUMMARY:
A longitudinal pilot study will be conducted to determine if there are additional testing modalities that are effective in broadly phenotyping subclinical dysfunction in patients with Fabry disease. Individual patients will undergo serial testing over a two-year period to evaluate for changes in their cardiovasculaorenal function during this period. Novel modalities evaluated will include measures of arterial stiffness, ambulatory blood pressure monitoring, cardiopulmonary exercise testing (CPET), and novel serum and urine biomarkers. The benefit of these measures being evaluated is that they are noninvasive, can be performed rapidly, and have reduced costs compared to the current standard screening modalities. Results from these evaluations will be compared to cMRI and standard urine and serum biomarkers performed clinically per local standard of care. The results will also be compared to both published normative data and data from patients with diabetes mellitus, who have a similar microvascular disease process to patients with Fabry disease.

ELIGIBILITY:
Inclusion Criteria:

* Fabry patients with classical disease
* English speaking, which is needed to assist with obtaining a maximal effort CPET
* No medical contraindications to cardiopulmonary exercise testing or cMRI
* Either treatment naïve or current taking ERT

Exclusion Criteria:

* Physical limitation that would preclude exercise
* Currently prescribed non-ERT treatments for Fabry disease

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants to be included in this study are patients who are being seen for follow up of known Fabry disease. These patients are screened regularly by the Department of Human Genetics for routine Fabry disease care. All Fabry disease patients who are physically able have a baseline cMRI and CPET performed at their appointment, per local standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Peak systolic blood pressure | through study completion, approximately 22 months
  The mean peak systolic blood pressure for Fabry disease patients is assumed to be 160 mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No